CLINICAL TRIAL: NCT01870232
Title: EVALUATION OF USE OF ULTRASOUND FOR GREATER PALATINE NERVE BLOCK AND INFERIOR ALVEOLAR NERVE BLOCKS: AN OPEN LABEL FEASIBILITY STUDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Sugantha Ganapathy, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103294
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Greater Palatine Nerve Block; Inferior Alveolar Nerve Block
Keywords: Greater palatine nerve Block; Inferior Alveolar nerve block; dental anesthesia; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- US guided block (Experimental): Greater palatine nerve or inferior alveolar nerve blocks will be performed under US guidance
  Interventions: Procedure: US guided block

INTERVENTIONS:
Procedure: US guided block — Greater palatine nerve or inferior alveolar nerve blocks will be performed under US guidance

SUMMARY:
Dental anesthesia is routinely performed based on anatomical landmarks which can be variable leading to repeated injections and failure. Ultrasonography can be used to guide these injections by identifying the nerves, accompanying blood vessels and the bony landmarks. 20 healthy adult patients will be selected to receive ultrasound guided greater palatine nerve block (gpn) (10 patients) or inferior alveolar nerve (ian) block (10 patients) depending on the dental procedure they are undergoing. The study will evaluate the feasibility and success rates of the ultrasound guided gpn and ian nerve block.

DETAILED DESCRIPTION:
The study will be done on 10 adult patients belonging to asa physical status 1 or 2 undergoing dental procedures with indications for greater palatine or inferior nerve blocks. The study will be conducted in the dental clinic, university hospital, london health sciences centre. All subjects will receive the letter of information at least 4-6 hours before the study procedure. One of the investigators will obtain an informed consent prior to the procedure. All subjects will be clinically examined to rule out any contraindications to the block such as infection, allergy to local anesthetic and any known coagulopathic disorder. No sedation will be used. The study subjects will be positioned on the dental chair and requested to open the mouth as wide as possible. In patients undergoing dental procedure to the upper teeth posterior to canine, a linear hockey stick probe will be positioned long axis to the palate just medial to the alveolar ridge. A color doppler will be used to identify the greater palatine artery (gpa) and this artery will be traced to the greater palatine (gpn) foramen by moving the probe gradually posteriorly until the greater palatine foramen is visualized and the gpn and the gpa are seen to exit from the foramen. Using an oblique off-plane approach a 25g needle attached to a dental carpule of 2% lidocaine will be inserted to contact the nerve and a total of 1ml of local anesthetic is deposited around the nerve and the needle removed. In patients undergoing a dental procedure in mandible, the ian block will be done with the same probe. The ultrasound probe will be positioned so that it is facing laterally on the buccal mucosa close the retromolar area. A color doppler will be used to identify the inferior alveolar artery and a 25g needle coming in-plane to the probe from the anterior side of the probe will deposit the local anesthetic agent perineurally. Images will be stored pre-injection, during injection and post injection. One of the investigators will test for the sensory block in the distribution of gpn and ian. The sensory anesthesia is graded as no anesthesia, partial anesthesia and complete anesthesia for each of the nerve blocks. The time to perform the blocks and time to block onset will also be noted. The total procedure duration is counted form the time of starting the scan to the time of completion of injection. The block performance duration is documented from the time of starting the needle insertion to the end of injection. Time from the end of injection to onset of sensory analgesia will be considered as the onset time. The blocks will be tested at 2 minutes, 5 minutes and 10 minutes after the injection. For the gpn, the sensory block will be documented on the hard palate from the last molar to the canine on the blocked side specifically at the 1st premolar mesially. The areas that will be tested with the dental probe for ian are the buccal mucosa at the base of the first molar tooth (ian), the lower lip of the blocked side, the tip of the tongue (lingual nerve) as well as the lingual mucosa (lingual nerve ) and the buccal mucosa lateral to the molars on the block side (ian). Occurrence of any local hematoma or paresthesia during the procedure will be documented. The subjects will be contacted over the telephone at 24 hours for any residual paresthesia or numbness.

ELIGIBILITY:
Inclusion Criteria:

1. MALE AND FEMALES PATIENTS
2. MANDIBULAR OR MAXILLARY DENTAL PROCEDURES IN THE DISTRIBUTION OF GREATER PALATINE OR INFERIOR ALVEOLAR NERVES.
3. ASA CLASS I, II

Exclusion Criteria:

1. ASA III AND IV
2. KNOWN NERVE INJURY OR NEUROPATHIES IN THE INTENDED BLOCK DISTRIBUTION
3. PATIENTS WITH KNOWN COAGULOPATHY
4. PATIENTS WITH KNOWN ALLERGY TO LOCAL ANESTHETIC OR THE PRESERVATIVE
5. PSYCHIATRIC ILLNESSES
6. LACK OF INFORMED CONSENT.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of nerve blocks | 10 minutes
  the success rate of the blocks will be tested at 2, 5 and 10 minutes following the ultrasound guided injections. no anesthesia at the end of 10 minutes will be termed block failure

CONTACTS AND LOCATIONS:
Overall Officials: Sugantha Ganapathy, FRCPC, Principal Investigator — Professor, Director, regional and Pain reseaerch
Locations (1):
- London Health Sciences Centre University Hospital, London, Ontario, Canada